Exploring the Effectiveness of the Intentionality the Matrix of Healing in Enhancing
Oral Health Education Outcomes for Community-Dwelling Middle-Aged and Older
Adults

## **Abstract**

Healthy aging is becoming increasingly important. As individuals age, three major symptoms—sarcopenia, dysphagia, and frailty—may develop. Early detection of oral functional decline and the implementation of oral health practices are essential for improving the quality of life in older adults. However, few studies have focused on the sustainability of self-care behaviors following oral health education among community-dwelling middle-aged and elderly individuals. Therefore, this study aims to apply the intentionality the matrix of healing framework as an intervention in community-based oral health education for middle-aged and elderly individuals to evaluate its effectiveness. A parallel randomized experimental design will be adopted, recruiting 90 middle-aged and elderly individuals from community through online channels. Participants will be randomly assigned to one of three groups: (1) Intentional interview combined with expressive arts activities, (2) Expressive arts activities only, or (3) Control group. Data on sarcopenia risk, eating assessment, grit, oral health literacy, and oral self-care behaviors were collected through questionnaires at baseline, one week after the intervention, and at a one-month follow-up. Statistical analyses, including descriptive statistics and inferential tests, were performed. The findings of this study are expected to provide evidence-based insights into the risks of sarcopenia and oral functional decline among community-dwelling older adults, while also offering empirical support for enhancing grit, oral health literacy, and oral selfcare behaviors. Ultimately, the results will contribute to advancing education, nursing practices, and policy development to improve the quality of life for middle-aged and elderly individuals in the community.

Keywords: Intentionality the matrix of healing; Community; Middle-aged and older adults; Oral health education

1

Version: 2; Date: 2025.5.16